CLINICAL TRIAL: NCT00053885
Title: A Phase II Study of PTK787/ZK222584 (NSC#719335) in Patients With Unresectable Malignant Mesothelioma
Brief Title: PTK787/ZK 222584 in Treating Patients With Unresectable Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-30107; U10CA031946 (NIH); CALGB-30107; CDR0000269537 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Malignant Mesothelioma
Keywords: advanced malignant mesothelioma; epithelial mesothelioma; recurrent malignant mesothelioma; sarcomatous mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — vatalanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PTK787/ZK 222584 (Experimental): Patients receive oral PTK787/ZK 222584 daily. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 2 months for 1 year, every 4 months for 1 year, and then every 6 months for 1 year.
  Interventions: Drug: PTK787/ZK 222584

INTERVENTIONS:
Drug: PTK787/ZK 222584 — oral

SUMMARY:
RATIONALE: PTK787/ZK 222584 may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

PURPOSE: Phase II trial to study the effectiveness of PTK787/ZK 222584 in treating patients with unresectable malignant mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of PTK787/ZK 222584, in terms of 3-month progression-free survival, in patients with malignant mesothelioma.
* Determine the response rate in patients treated with this drug.
* Determine the toxicity of this drug in these patients.
* Determine the overall and failure-free survival of patients treated with this drug.
* Correlate pretreatment circulating serum levels of vascular endothelial growth factor (VEGF), platelet-derived growth factor, and VEGF mRNA isoforms with response in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral PTK787/ZK 222584 daily. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 1 year, every 4 months for 1 year, and then every 6 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant mesothelioma of 1 of the following types:

  * Epithelial
  * Sarcomatoid
  * Mixed
* Not amenable to radiotherapy or curative surgery
* Any site of origin including, but not limited to, the following:

  * Pleura
  * Peritoneum
  * Pericardium
  * Tunica vaginalis
* At least one unidimensionally measurable lesion outside of prior irradiation port

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * The following are not considered measurable:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 2.5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN
* Negative for proteinuria by dipstick OR
* Urinary protein no greater than 500 mg and creatinine clearance at least 50 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-barrier contraception
* No currently active second malignancy except non-melanoma skin cancers (unless therapy is completed and risk of relapse is less than 30%)
* No other concurrent uncontrolled illness
* No ongoing active infections
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior signal transduction inhibitor therapy
* No prior angiogenesis inhibitor therapy

Chemotherapy

* No prior cytotoxic chemotherapy for this malignancy
* No concurrent chemotherapeutic agents
* Prior intrapleural cytotoxic or sclerosing therapy (including bleomycin) allowed

Endocrine therapy

* No concurrent hormonal therapy except steroids for adrenal failure or hormones for non-disease-related conditions (e.g., insulin for diabetes)

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent palliative radiotherapy

Surgery

* See Disease Characteristics
* At least 2 weeks since prior major surgery

Other

* At least 30 days since prior investigational agents
* At least 7 days since prior grapefruit or grapefruit juice
* At least 7 days since prior CYP3A4 inducers
* No prior PTK787/ZK 222584
* No prior tyrosine kinase inhibitor therapy
* No other concurrent investigational agents
* No concurrent isoenzyme inducers or inhibitors of p450
* No concurrent warfarin or similar oral anticoagulants

  * Heparin allowed
* No concurrent grapefruit or grapefruit juice
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2003-07; Primary Completion 2005-07 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Survival | Up to 3 years post-treatment
Failure free survival | Up to 3 years post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Jahan, MD, Study Chair — University of California, San Francisco
Locations (80):
- United States (80):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Cancer Center at Memorial Regional Hospital, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at the Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - NorthEast Oncology Associates - Concord, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Comprehensive Cancer Center at Moore Regional Hospital, Pinehurst, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - University of Tennessee Cancer Institute at Methodist Central Hospital, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Incorporated - Roanoke, Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Result] Jahan TM, Gu L, Wang X, et al.: Vatalanib (V) for patients with previously untreated advanced malignant mesothelioma (MM): A phase II study by the Cancer and Leukemia Group B (CALGB 30107). [Abstract] J Clin Oncol 24 (Suppl 18): A-7081, 2006.
- [Derived] Jahan T, Gu L, Kratzke R, Dudek A, Otterson GA, Wang X, Green M, Vokes EE, Kindler HL. Vatalanib in malignant mesothelioma: a phase II trial by the Cancer and Leukemia Group B (CALGB 30107). Lung Cancer. 2012 Jun;76(3):393-6. doi: 10.1016/j.lungcan.2011.11.014. Epub 2011 Dec 22. PMID 22197613